CLINICAL TRIAL: NCT05445713
Title: A Cross-sectional, Observational Study to Characterise Long-COVID in an Urban Sample of South African Adults
Brief Title: A Cross-sectional, Observational Study to Characterise Long COVID-19 in an Urban Sample of South African Adults
Acronym: ChaLOC
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Professor Francois Venter, Professor, University of Witwatersrand, South Africa
Other Study IDs: EZ-FV-028
Record Dates: First submitted 2022-07-04; First posted 2022-07-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Full blood count: red cell count, haemoglobin, haematocrit, mean cellular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), red cell distribution width (RDW), white cell count and differential (neutrophil count, lymphocyte count, monocyte count, eosinophil count, and basophil count), and platelet count
  Liver function: total protein, albumin, total bilirubin, direct bilirubin, alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactate dehydrogenase (LDH)
  Renal function: urea, creatinine, estimated creatinine clearance (Cockcroft-Gault method), cystatin C
  DNA extraction for genotyping and sequencing at the Sydney Brenner Institute for Molecular Bioscience (SBIMB)
  Additional blood (50 mL) and urine (100 mL) samples will be stored for possible future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Asymptomatic subjects found to be PCR/antigen/antibody-positive during routine screening for SARS-CoV-2 infection
- Cohort 2: Symptomatic outpatients who were confirmed to have COVID-19 through a positive PCR/antigen test
- Cohort 3: Inpatients surviving hospitalisation for severe COVID-19 and who were PCR/antigen-positive
- Cohort 4: Participants vaccinated in clinical trials in 2020 prior to widespread community exposure, and hence protected from severe COVID-19 (and possibly Long-COVID) if subsequently infected.

SUMMARY:
"Long-COVID'' (also known as post-COVID-19 syndrome, post-acute sequelae of COVID-19, or chronic COVID syndrome, used here as 'Long-COVID' for brevity), is a complex array of postconvalescence symptoms following SARS-CoV-2 infection. The syndrome, common in COVID-19 survivors, can affect every organ system through as-yet uncharacterised but presumed immunological mechanisms. Prevalence depends on the definition used and time-period of follow-up, as well as the population being studied. The syndrome has been associated with significant and persistent disability in some survivors but has been hampered, until recently, by lack of a clinical definition, diagnostic criteria, and objective measures of disease or disability [1]. A Delphi-informed initial World Health Organisation (WHO) clinical definition was released in early October 2021 but has attracted much criticism from both clinicians and survivors for a host of reasons, ranging from a lack of precision to a lack of inclusion [2].

Further complicating the syndrome is the context in which the SARS-CoV-2 epidemic occurred, which was associated with severe lockdowns in many countries (including South Africa) with social isolation, widespread fear and disinformation, widespread economic hardship, and loss of family and acquaintances, all of which contribute to symptoms (psychiatric and sleep disturbances, pain, and other syndromes) reported to be associated with Long-COVID. Finally, many Long-COVID symptoms overlap with those seen in patients hospitalised for any severe illness, especially those admitted to intensive care and ventilated. However, the proliferation of literature reporting associations of Long-COVID symptoms with more severe COVID-19 disease, and objective immunological, radiological, and organ-specific dysfunction in those reporting symptoms, suggests that the entity is real. The pathogenesis of Long-COVID is poorly understood, but this association with more severe disease - where immune dysregulation plays a major role in those with hospitalization, respiratory failure, and death - suggests an immune-mediated inflammatory dysfunction that may impact all organs [3-14].

The sheer rapidity of four major infection waves in South Africa, the initial focus on containing the hospital burden of those with severe illness, and subsequent emphasis on the roll-out of a mass vaccination program, has left little space for studying SARS-COV-2 sequalae in survivors. This group, loosely and inaccurately termed "recovered'' in South African reporting, were largely unvaccinated or partly vaccinated at the time of infection, leaving them at risk of developing Long-COVID.

DETAILED DESCRIPTION:
This is a single-centre, follow-up, observational, cross-sectional study of four distinct, longitudinal cohorts. Extensive clinical history will be obtained from each participant, and symptom questionnaire characterisation of Long-COVID (with a strong focus on organ-specific dysfunction, psychiatric, sleep, and pain parameters - all of which appear to be major features of Long-COVID), as well as laboratory and genetic characterisation will be performed. A subset of each cohort will be randomly selected for more specific syndrome characterisation related to sleep and pain, respiratory, cardiology, renal and glucose metabolism.

The consequences of Long-COVID will be described and compared in four large, well-described clinical cohorts of African patients surviving SARS-CoV-2:

* Cohort 1: asymptomatic subjects found to be PCR/antigen/antibody-positive during routine screening for SARS-CoV-2 infection
* Cohort 2: symptomatic outpatients who were confirmed to have COVID-19 through a positive PCR/antigen test
* Cohort 3: inpatients surviving hospitalisation for severe COVID-19 and who were PCR/antigen-positive
* Cohort 4: participants vaccinated in clinical trials in 2020 prior to widespread community exposure, and hence protected from severe COVID-19 (and possibly Long-COVID) if subsequently infected.

After obtaining informed consent from potential participants, a single cross-sectional, baseline visit will be conducted for each participant. Demographic data, clinical history (including COVID-19 history, targeted symptoms, and risk factors), COVID-19 vaccination dates (if administered), and details of previous and concomitant medications will be collected. Multiple questionnaires related to psychiatric screening, psychosocial factors, work function assessment, sleep quality, and pain assessment will be administered. Respiratory and cardiac function will be evaluated through a dyspnoea scale, walking test and an ECG. Laboratory evaluations will include a full blood count, serum chemistry, liver function tests, renal function assessment, inflammatory markers, and DNA extraction for genotyping. Blood and urine samples will be stored locally for possible future analysis. Human immunodeficiency virus (HIV) testing will be performed for participants consenting to this optional assessment.

After the baseline visit, participants with Long-COVID will be identified using the WHO clinical definition and general health assessments [2]. Randomly selected sub-groups of participants with, and without, Long-COVID will be selected from each of the four cohorts for additional investigations through participation in the following sub-studies:

* Respiratory evaluation: dyspnoea assessment, high-resolution computed tomography (CT) scan, lung function studies including spirometry and diffusion capacity (DLCO) [Section 7.2.2.1]
* Cardiac evaluation: clinical history and examination, serial blood pressure, six minute walk test (distance), ECG, echocardiogram including speckle tracking, cardiac magnetic resonance imaging (MRI), creatine kinase MB fraction (CK-MB), cardiac troponin T (cTnT), prohormone brain natriuretic peptide (pro-BNP), and possible coronary angiography in patients with acute coronary syndromes and unstable angina [Section 7.2.2.2]
* Psychiatric and neuroendocrine evaluation: questionnaires/surveys, semi-structured interview, home visit, saliva cortisol analysis, collection of diary data, actigraphy, adrenocorticotropic hormone (ACTH) challenge (cosyntropin sensitivity test [CST]), cellular immunity assessment [Section 7.2.2.3]
* Sleep evaluation: questionnaires, actigraphy with sleep diaries, polysomnography (PSN) [Section 7.2.2.4]
* Pain evaluation: quantitative sensory testing (QST) and conditioned pain modulation (CPM) assessments [Section 7.2.2.5]
* Glucose metabolism evaluation: oral glucose tolerance test (OGTT) including assessment of glucose, insulin, and c-peptide to estimate insulin sensitivity and beta-cell function [16]. [Section 7.2.2.6] Abnormalities detected in the assessments (including undiagnosed mental health issues) will be managed by on-study medical personnel with referral as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written or electronic informed consent for the baseline visit prior to any study-specific assessment or procedure.
2. Age at least 18 years at the time of signing the informed consent form.
3. Previous asymptomatic SARS-CoV-2 infection, confirmed through a documented positive PCR, antigen, or antibody test, at least six months prior to the baseline visit [Cohort 1 only] or, previous symptomatic SARS-CoV-2 infection for which hospitalisation was not required, confirmed through a documented positive PCR or antigen test at the time, at least six months prior to the baseline visit [Cohort 2 only] or, previous hospitalisation for management and treatment of COVID-19 confirmed through a documented positive PCR or antigen test at the time, at least six months prior to the baseline visit [Cohort 3 only] or, previous asymptomatic or symptomatic SARS-CoV-2 infection, confirmed through a documented positive PCR, antigen, or antibody test, at least six months prior to the baseline visit and received a COVID-19 vaccine in a non-placebo arm of a COVID-19 vaccine study during 2020 [Cohort 4 only].
4. Willing to consent to verification of vaccination status on the national Electronic Vaccination Data System (EVDS).
5. Access to a reliable telephone or other device permitting information transfer.

Exclusion Criteria:

1. Symptomatic SARS-CoV-2 infection at any stage prior to the baseline visit [Cohort 1 only].
2. SARS-CoV-2 infection, confirmed through a documented positive PCR, antigen, or antibody test, prior to vaccination in a non-placebo arm of a COVID-19 vaccine study during 2020 [Cohort 4 only].
3. COVID-19 within three months of the baseline visit.
4. Personnel (e.g., investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study.
5. Any physical, mental, or social condition, that, in the Investigator's judgment, might interfere with the completion of the baseline assessments and evaluations. The Investigator should make this determination in consideration of the volunteer's medical history.
6. Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults at least 18 years of age with previous confirmed SARS-CoV-2 infection (symptomatic or asymptomatic) will be invited to participate. Approximately 400 participants will be enrolled.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
To characterise Long-COVID in four cohorts of patients | 6 Months
  Incidence, severity, and duration of Long-COVID symptoms.

SECONDARY OUTCOMES:
Inflammatory markers | 6 Months
  High sensitivity C-reactive protein (hs-CRP)
Inflammatory markers | 6 Months
  Interleukin-1
Inflammatory markers | 6 Months
  Interleukin-6 (IL-6)
Inflammatory markers | 6 Months
  Interleukin-8 (IL-8)
Inflammatory markers | 6 Months
  Tumour necrosis factor alpha
Inflammatory markers | 6 Months
  Tumour necrosis factor alpha receptor-1 (TNFR1)
Inflammatory markers | 6 Months
  Monocyte chemoattractant protein-1 (MCP-1)
Psychological profiles | 6 Months
  Headache Impact Test-6
Psychological profiles | 6 Months
  Patient Health Questionnaire-9
Psychological profiles | 6 Months
  Generalised Anxiety Disorder 7
Psychological profiles | 6 Months
  PTSD Checklist for DSM-5 - Civilian Version
Psychological profiles | 6 Months
  Mood Disorder Questionnaire; a short screening tool evaluating the symptoms of bipolar disorder
Psychological profiles | 6 Months
  Montreal Cognitive Assessment
Psychological profiles | 6 Months
  Daily Fatigue Impact Scale; a survey tool that assesses physical, cognitive, and psychosocial dimensions of fatigue in everyday life
Psychosocial exposures | 6 months
  COVID-19 related stress questionnaire
Psychosocial exposures | 6 months
  Multidimensional Scale of Perceived Social Support; a brief research tool designed to measure perceptions of support from 3 sources - family, friends, and a significant other; the scale is comprised of a total of 12 items, with 4 items for each subscale
Psychosocial exposures | 6 months
  Perceived Stress Scale
Psychosocial exposures | 6 months
  Adverse Childhood Experiences tool
Work performance in employed participants | 6 months
  Normal activities and work productivity questionnaire; daily diaries
Sleep quality and disorders | 6 months
  Pittsburgh Sleep Quality Index
Sleep quality and disorders | 6 months
  Epworth Sleepiness Scale
Sleep quality and disorders | 6 months
  Berlin Questionnaire for risk of sleep apnoea
Sleep quality and disorders | 6 months
  International Restless Legs Syndrome Severity Scale
Sleep quality and disorders | 6 months
  Sleep quality and mood visual analogue scale
Pain experience | 6 months
  Brief Pain Inventory
Cardiorespiratory function | 6 months
  Modified Medical Research Council Dyspnoea Scale
Cardiorespiratory function | 6 months
  Six-minute walk test (distance)
Cardiorespiratory function | 6 months
  ECG parameters and morphology
Standard laboratory parameters | 6 months
  Full blood count
Standard laboratory parameters | 6 months
  Serum chemistry
Standard laboratory parameters | 6 months
  Liver function tests
Standard laboratory parameters | 6 months
  Glucose, HbA1C
Renal function | 6 months
  Creatinine clearance
Renal function | 6 months
  Cystatin-C
Renal function | 6 months
  Urine dipstick parameters
Renal function | 6 months
  Urine albumin-to-creatinine ratio
Host genetic factors that may be associated with Long-COVID | 6 months
  Genotyping results
Host genetic factors that may be associated with Long-COVID | 6 months
  DNA sequencing results

CONTACTS AND LOCATIONS:
Overall Officials: Francois WD Venter, MBBCh, Principal Investigator — Ezintsha, a division of Wits Health Consortium; Simiso M Sokhela, MBBCh, Study Director — Ezintsha, a division of Wits Health Consortium; Nonkululeko Mashabane, BPharm, Study Chair — Ezintsha, a division of Wits Health Consortium
Locations (2):
- South Africa (2):
  - Sunnyside Office Park, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital (CMJAH), Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data

DOCUMENTS (2):
  • Study Protocol (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05445713/Prot_000.pdf
  • Informed Consent Form (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT05445713/ICF_001.pdf